CLINICAL TRIAL: NCT07295132
Title: A Randomized Clinical Trial Evaluating the Role of Secondary Cytoreductive Surgery Following Neoadjuvant Chemotherapy in Platinum-Sensitive Recurrent Ovarian Cancer: Patient Selection Informed by CA-125 Response Dynamics During Chemotherapy (RESCUE Study)
Brief Title: RESCUE Study (REcurrent Ovarian Cancer Secondary Cytoreduction Using Chemotherapy rEsponse)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korean Gynecologic Oncology Group (Other)
Responsible Party: Principal Investigator, Dae-Yeon Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS-2025-02273048; RS-2025-02273048 (Other Grant/Funding Number: Korea Health Industry Development Institute(KHIDI))
Record Dates: First submitted 2025-11-18; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer Recurrent; Platinum Sensitive Ovarian Cancer
Keywords: platinum sensitive recurrent ovarian cancer; secondary cytoreductive surgery; neoadjuvant chemotherapy; CA-125 response
MeSH Terms: interventions — Platinum Compounds

STUDY DESIGN:
Intervention Model Description: In this study, following neoadjuvant chemotherapy, patients are randomized to one of two arms: either receiving Secondary Cytoreductive Surgery followed by the remaining chemotherapy, or continuing with chemotherapy alone, in order to evaluate which strategy leads to superior Progression-Free Survival.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Experimental): Neoadjuvant platinum-based chemotherapy and Secondary cytoreductive surgery followed by the remaining chemotherapy
  Interventions: Procedure: Secondary cytoreductive surgery; Drug: Platinum Based Chemotherapy
- No surgery (Active Comparator): platinum-based chemotherapy
  Interventions: Drug: Platinum Based Chemotherapy

INTERVENTIONS:
Procedure: Secondary cytoreductive surgery — Secondary Cytoreductive Surgery (SCS) is a surgical procedure performed on patients with relapsed or recurrent epithelial ovarian cancer, after they have completed their initial course of treatment (such as primary surgery and chemotherapy).
  Arms: Surgery
Drug: Platinum Based Chemotherapy — Platinum Based Chemotherapy

SUMMARY:
This is a multicenter, prospective, randomized, open-label Phase III clinical trial (RESCUE study) evaluating the efficacy of secondary cytoreductive surgery (SCS) in patients with platinum-sensitive recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer who have shown a favorable response to 3-4 cycles of platinum-based neoadjuvant chemotherapy and are assessed as highly likely to achieve complete tumor resection based on selection models. Eligible patients will be randomly assigned to either the experimental arm, receiving SCS followed by chemotherapy (with or without maintenance), or the active comparator arm, receiving chemotherapy only (with or without maintenance), with the primary objective being to compare the Progression-Free Survival (PFS) between the two groups to determine the additional clinical benefit of SCS in this carefully selected patient population.

DETAILED DESCRIPTION:
The RESCUE study is a major clinical trial focused on improving treatment for women battling recurrent ovarian, fallopian tube, or primary peritoneal cancer. These cancers, which often return after initial treatment, are known to be aggressive. The challenge for doctors is deciding when and if a second major surgery, known as secondary cytoreductive surgery (SCS), will truly benefit the patient.

The Study's Focus: When is Surgery Best?

Currently, when the cancer returns, patients receive chemotherapy. The key question is whether adding a challenging surgery (SCS) to the chemotherapy offers better survival chances than chemotherapy alone. Past studies have suggested that SCS is only helpful if the surgeon can remove all visible signs of cancer.

The RESCUE study addresses this by using a modern, personalized approach:

Selection: The study enrolls patients whose cancer is platinum-sensitive (meaning it responded well to the initial platinum-based chemotherapy).

Pre-Surgical Test: Patients first receive several cycles of chemotherapy. During this time, the research team uses a special model to analyze how quickly a tumor marker called CA-125 decreases. This dynamic change in the marker helps doctors predict, with greater accuracy than ever before, which patients are most likely to achieve a complete resection (removal of all visible disease) during surgery.

Randomization: Patients who are identified as strong candidates for complete resection are then randomly assigned (like flipping a coin) into one of two groups:

Group 1 (Experimental): Receive the carefully planned secondary cytoreductive surgery followed by the rest of their chemotherapy.

Group 2 (Control): Continue with chemotherapy alone, without the surgery.

The Goal

The primary goal of the RESCUE study is to determine if adding secondary cytoreductive surgery provides a significant advantage in Progression-Free Survival (PFS)-the length of time a patient lives without their cancer getting worse-for this highly selected group of patients.

By meticulously selecting the patients most likely to benefit from surgery, this trial aims to establish a new standard of care, ensuring that this major surgical procedure is performed only when it is expected to yield the best possible outcome for the patient.

ELIGIBILITY:
Inclusion Criteria:

* First recurrence of platinum-sensitive, invasive epithelial ovarian, fallopian tube, or primary peritoneal cancer, regardless of initial stage.
* A progression-free interval of at least 6 months after the end of the last platinum-containing regimen.
* Demonstrated response during neoadjuvant chemotherapy after recurrence (Complete Response/Partial Response/Stable Disease according to RECIST 1.1 or GCIG CA-125 response, which is a ≥50% reduction in pre-treatment CA-125 level sustained for ≥28 days).
* Women aged 19 years or older.
* The tumor is judged to be completely resectable by surgery (R0) based on the judgment of an experienced surgeon
* Patients who provide signed and written informed consent and consent to data transfer and processing.

Exclusion Criteria:

* Patients without recurrence
* Patients with non-epithelial tumors or borderline tumors.
* Patients with second, third, or subsequent recurrence.
* Patients with a secondary malignancy treated with laparotomy and other neoplasms, where the treatment is expected to interfere with the treatment of recurrent ovarian cancer or significantly affect prognosis.
* Patients with platinum-refractory tumors (i.e., progression during chemotherapy or recurrence within 6 months after the end of the previous first platinum-containing regimen).
* Cases where only palliative surgery is planned.
* Radiological signs suggestive of metastasis that are considered completely unresectable.
* Any comorbidity that precludes surgery and/or chemotherapy (e.g., poor general condition, severe infection, conditions that may cause severe bleeding, severe renal disease, etc.).
* Any medical history that may cause excessive surgical risk pre- or post-operatively.
* Medications being taken that pose a significant surgical risk (e.g., oral anticoagulants, bleeding risk due to bevacizumab).
* Absence of evaluable archived tumor tissue.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The length of time a patient lives with a cancer, without the disease getting worse or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  the date of randomization into the study arm until the date of death from any cause
Complete Resection Rate (R0) | postoperative (up to 2 months after surgery)
  The Complete Resection Rate is the percentage of patients in the surgical arm for whom the surgeon successfully removes all macroscopic (visible) tumor tissue (R0 status).
Surgical Complication Rate | Postoperative (up to 2 months after surgery)
  The Surgical Complication Rate measures the frequency and severity of adverse events, such as infections, bleeding, or wound healing problems (graded by Clavien-Dindo classification), experienced by patients in the Secondary Cytoreductive Surgery arm.
KELIM (The modeled CA-125 ELIMination rate constant K) | Baseline
  The KELIM (The modeled CA-125 ELIMination rate constant K) Score will be evaluated as a secondary endpoint to confirm its prognostic accuracy in predicting the actual surgical outcome (Complete Resection Rate) and the long-term survival (PFS and OS) in the randomized patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Yeon Kim, Principal Investigator — Asam Medical Center

IPD SHARING:
Plan to Share IPD: Undecided